CLINICAL TRIAL: NCT01764971
Title: Cerebral Dysfunction in Chronic ITP With High Risk of Serious Bleeding Excluding Intracranial Hemorrhage.
Brief Title: Cerebral Dysfunction in Chronic ITPwith High Risk of Serious Bleeding Excluding Intracranial Hemorrhage.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professor of pediatrics, Ain Shams University
Other Study IDs: CNS and chronic ITP
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Thrombocytopenia
Keywords: Chronic ITP, Cerebral dysfunction
MeSH Terms: interventions — Wechsler Scales; Wisconsin Card Sorting Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- chronic itp and cerebral dysfunction: patients with chronic itp and had behavioral and or cognitive dysfunction
  Interventions: Other: IQ assessment and visual- motor assessment; Other: EEG,brain imaging
- chronic itp only: chronic ITP patients without cerebral dysfunction
  Interventions: Other: IQ assessment and visual- motor assessment

INTERVENTIONS:
Other: IQ assessment and visual- motor assessment — Psychological examination and evaluation for both groups to diagnose those with behavioral and /or cognitive dysfunction.
  Other Names: Benton visual retention test (BVRT); Wechsler Intelligence Scale; Wisconsin Card Sorting test
Other: EEG,brain imaging — For patients with cognitive or behavioral deficit, MRI brain and quantitative EEG will be done to identify any CNS abnormality.
  Other Names: quantitative EEG; MRI brain
  Groups: chronic itp and cerebral dysfunction

SUMMARY:
Intracranial hemorrhage despite being rare, several chronic ITP patients experience moderate to severe behavioral problems including learning difficulties, memory affection .These changes could be due to the presence of minute capillary dysfunction

DETAILED DESCRIPTION:
* First identify the presence of cognitive, behavioral and/or minimal neurological deficit in patients with chronic ITP and correlate these changes with radiological evidence of minimal CNS bleeding.
* Second investigate the correlation between these behavioral and/or minimal neurological deficits and duration, site and severity of bleeding (a total of 200 patient of persistently low platelet count < 20x 10 9 for at least more than one month duration).
* The aim is to assess the behavioral changes in chronic ITP patients, and to assess the possible relation of such changes to duration and recurrence of very low platelet count as well as pattern of bleeding excluding frank intracranial hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic ITP patients with persistent platelet count < 20 x 109/L for a period more than one month.
2. Chronic ITP with more than one attack of wet purpura and OR internal bleeding.

Exclusion Criteria:

1. Patients' with platelet count persistently more than 40 x 109/L.
2. Past history of intracranial hemorrhage.
3. Past history of known neurological or psychological deficit diagnosed before onset of ITP diagnosis

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from those treated in Hematology Clinic, Ain Shams University.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
cognitive, behavioral and/or minimal neurological deficit in patients with chronic ITP | 6 month
  cognitive, behavioral and/or minimal neurological deficit in patients with chronic ITP and correlate these changes with radiological evidence of minimal CNS bleeding.

SECONDARY OUTCOMES:
duration, site and severity of bleeding effect of duration, site and severity of bleeding | 6 months
  behavioral and/or minimal neurological deficits and duration, site and severity of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S Elalfy, professor, Principal Investigator — Ain Shams University
Locations (1):
- hematology clinic, pediatric hospital, Ain Shams University, Cairo, Egypt